CLINICAL TRIAL: NCT04146155
Title: Liraglutide Efficacy and Action on Type 2 Diabetes With Peripheral Atherosclerotic intErmittent Claudication (LEADPACE STUDY): a Prospective, 24-week, Multicenter, Randomized, Controlled Clinical Study
Brief Title: Efficacy and Safety of Liraglutide in Type 2 Diabetes With Lower Extremity Arterial Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zhengchao
Record Dates: First submitted 2019-10-16; First posted 2019-10-31 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes; Peripheral Vascular Disorder Due to Diabetes Mellitus
Keywords: Glucagon-like peptide-1; Claudication; Peripheral vascular disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Claudication; Peripheral Vascular Diseases | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide+standard-of-care treatment (Experimental): Intervention: Liraglutide is added to existing standard-of-care treatment containing one or more oral anti-hyperglycemic agents or insulin or a combination of these agents with the exception of other incretin and SGLT2i therapies.
  Interventions: Drug: Liraglutide+standard-of-care treatment
- standard-of-care treatment (Active Comparator): standard-of-care treatment with the exception of incretin and SGLT2i therapies. This approach expect to yield similar glycemic control in the two study groups.
  Interventions: Other: standard-of-care treatment

INTERVENTIONS:
Drug: Liraglutide+standard-of-care treatment — Liraglutide is available if pre-filled pens (6 mg/ml) as a solution for injection (Victoza®). One ml of solution contains 6 mg of Liraglutide (human glucagon-like peptide-1 analogue produced by recombinant DNA technology in Saccharomyces cerevisiae). One pre-filled pen contains 18 mg Liraglutide in 3 ml.
  Liraglutide is added to existing standard-of-care treatment containing one or more oral anti-hyperglycemic agents or insulin or a combination of these agents with the exception of other incretin and SGLT2i therapies in accordance with local clinical practice guidelines.
  Other Names: Victoza
  Arms: Liraglutide+standard-of-care treatment
Other: standard-of-care treatment — Standard-of-care treatment including: metformin should be given as the first line therapy as long as it is tolerated and not contraindicated; other agents, including sulfonylureas or glucosidase inhibitor or insulin, should be added to metformin .Glycemic control will be managed by the investigators in accordance with local clinical practice guidelines by the adjustment of concomitant glucose-lowering agents or the addition of new antidiabetic medications with the exception of incretin and SGLT2i therapies. This approach expect to yield similar glycemic control in the two study groups.
  Arms: standard-of-care treatment

SUMMARY:
Diabetic lower extremity arterial disease ( DLEAD ), is a common complication of type 2 diabetes. However, DLEAD remains less studied than other diabetic vascular complications; and only few randomised controlled trials (RCTs) have dealt with major lower-limb adverse events as prespecified endpoints. Studies have suggested that glucagon-like peptide-1 (GLP-1) analogues have a protective effect on the development of atherosclerosis, potentially mediated via the GLP-1 receptors expressed on endothelial cells, smooth muscle cells, and in monocytes/macrophages. The investigators aim to evaluate the improvement of lower extremity ischemia in patients with type 2 diabetes mellitus complicated with lower limb vascular lesions after liraglutide, compared with the standard-of-care treatment group.

DETAILED DESCRIPTION:
GLP-1 is an incretin hormone that mediates glucose-stimulated insulin secretion.Accumulating data from both animal and human studies confirmed a beneficial effect of GLP-1 on myocardium, endothelium and vasculature, suggesting the potential ameliorative effect of peripheral atherosclerosis. In our preliminary studies shown that liraglutide, a long-acting GLP-1R agonist (GLP1RA), stimulate endothelial proliferation and angiogenesis. The study aims to test the hypothesis that sustained activation of the GLP-1R enhances microvascular perfusion, promotes angiogenesis, leading to increased walking distance and limb perfusion in diabetes patients with peripheral arterial disease (PAD). Eligible patients will be randomized 1:1 to with or without liraglutide treatment by a 6-month follow-up. The primary endpoints are the change in initial and absolute claudication distance and assessment of limb ischemia at 6 months compared with baseline. This trial will collect important mechanistic and clinical information on the safety and efficacy of liraglutide in T2DM patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* type 2 diabetes (1999 WHO criteria)
* 7.5≤HbA1c ≤14%
* Age > 40 years
* lower extremity PAD with symptom
* Absence of distal arterial pulse.
* ABI less than 0.9 or the value decreased by more than 15% after treadmill test.
* Presence of stenosis or occlusion of lower extremity arteries as determined by Duplex ultrasound imaging or lower extremity CTA; or lower extremity DSA(Digital Substraction Angiography).

Exclusion Criteria:

* Type 1 diabetes
* Other Concomitant illness:

  1) poorly controlled hypertension: >160 mmHg systolic blood pressure and/or>100 mmHg diastolic blood pressure (with or without long-term oral antihypertensive drugs); 2) Chronic heart failure NYHA class (III-IV); 3) An acute coronary or cerebro-vascular event within the previous 6 months; 4) hematological malignancies such as acute or chronic myeloid leukemia, or any other hematological disorders that would interfere with the determination of circulating EPC levels; 5) Personal history of non-familial medullary thyroid carcinoma; 6) Immunological disorders such as lupus, psoriasis, scleroderma and rheumatoid arthritis which would interfere with the determination of circulating EPC levels; 7) Chronic haemodialysis or chronic peritoneal dialysis; 8) End stage liver disease, presence of acute or chronic liver disease or recent history of the following: ALT level ≥ 3 times the upper limit of normal, or AST level ≥ 3 times the upper limit of normal; 9) Severe gastrointestinal diseases, such as gastrointestinal ulcer, gastrointestinal bleeding, pyloric stenosis, gastric bypass surgery; 10) History of chronic pancreatitis or idiopathic acute pancreatitis; 11) Any acute condition or exacerbation of chronic condition that would in the Investigator's opinion interfere with the initial trial visit schedule and procedures; 12) Inability to walk on a tredamill without grade at a speed of at least 3.2 km/h for at least 2 minutes.
* Drugs: 1) Known or suspected hypersensitivity to trial products or related products ; 2) Use of GLP-1 receptor agonist (exenatide (BID or OW), liraglutide, or other) within 6 months prior to screening; 3).Alcohol or drugs abuse.
* 4. Acute decompensation of glycaemic control requiring immediate intensification of treatment to prevent acute complications of diabetes (eg diabetes ketoacidosis) within 90 days prior to screening.
* Recent (within 6 months) surgery or trauma.
* Pregnancy and lactation.
* Psychiatric disorders
* Simultaneous participation in any other clinical trial of an investigational agent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Initial and absolute claudication distance | 24 weeks
  The primary outcome measures used to assess efficacy were pain-free walking distance (distance walked to the onset of symptoms, or the initial claudication distance [ICD]) and the maximum distance walked (absolute claudication distance [ACD]) on standardized treadmill testing. Evaluation of walking performance was accomplished with standardized treadmill testing. A constant speed of 3.2 km/h (2mile/h) and a fixed incline of 12.5% were used.

SECONDARY OUTCOMES:
Assess the effects on ABI of a six month treatment with Liraglutide compared to control group (standard-of-care treatment). | 24 weeks
  ankle-brachial index is ratio of ankle systolic pressure to arm systolic pressure: using a 10-12 cm sphygmomanometer cuff placed just above the ankle and a doppler instrument used to measure the systolic pressure of the posterior tibial and dorsalis pedis arteries of each leg. These pressures are then normalized to the higher brachial pressure of either arm to form the ankle-brachial index (ABI). The index leg is often defined as the leg with the lower ABI.
Assess the effects on endothelial function of a six month treatment with Liraglutide compared to control group (standard-of-care treatment). | 24 weeks
  Assess the effects on endothelial function of a six month treatment with Liraglutide compared to conventional treatment, assessed as the baseline corrected change in endothelial function by flow-mediated vasodilation (FMD) of the brachial artery at 6 months.
Muscle microvascular perfusion by CEU | 24 weeks
  Contrast enhanced ultrasound (CEU) performed by experienced radiologists is used for contrast ultrasonographic examination of skeletal muscle.
Assess the effects on the endothelial circulating progenitor cells concentration of a six month treatment with Liraglutide compared to control group (standard-of-care treatment). | 24 weeks
  Circulating progenitor cells (EPCs) will be quantified using flow cytometry before and after 6 month treatment GLP-1 receptor agonist or conventional therapy (control group). Briefly, after erythrocyte lysis, peripheral blood will be stained with 10µL fluorescein isothiocyanate-conjugated anti-human CD34 mAb, 10µL phycoethrin-conjugated anti-human KDR mAb, and 10µL allophycocyanin-conjugated anti-CD133 mAb.
Changes from baseline in HbA1c | 24 weeks
  Change from baseline to last assessment during the treatment period in HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Chao Zheng, MD,PhD, Principal Investigator — the Second Affiliated Hospital Zhejiang University Schoolof Medicine; Youjin Pan, MD., Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Xia Li, MD,PhD, Principal Investigator — Central South University; Li Li, MD., Principal Investigator — Ningbo Hospital of Zhejiang University
Locations (1):
- The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kanie T, Mizuno A, Takaoka Y, Suzuki T, Yoneoka D, Nishikawa Y, Tam WWS, Morze J, Rynkiewicz A, Xin Y, Wu O, Providencia R, Kwong JS. Dipeptidyl peptidase-4 inhibitors, glucagon-like peptide 1 receptor agonists and sodium-glucose co-transporter-2 inhibitors for people with cardiovascular disease: a network meta-analysis. Cochrane Database Syst Rev. 2021 Oct 25;10(10):CD013650. doi: 10.1002/14651858.CD013650.pub2. PMID 34693515